CLINICAL TRIAL: NCT03258099
Title: Association of Genetic Polymorphisms With Capecitabine-based Chemotherapy Toxicities in Chinese Solid Tumor Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2016[1239]-1
Record Dates: First submitted 2017-08-17; First posted 2017-08-23 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumor; Capecitabine; Drug-Related Side Effects and Adverse Reactions; Pharmacogenetics; Pharmacokinetics
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wild genotype: Through next generation sequencing, distinguish wild genotype of capecitabine
  Interventions: Genetic: detection of genotype
- mutant genotype: Through next generation sequencing, distinguish mutant genotype of capecitabine
  Interventions: Genetic: detection of genotype

INTERVENTIONS:
Genetic: detection of genotype — detection of genotype by next generation sequencing

SUMMARY:
Capecitabine is one of the most active agents in the treatment of many kinds of solid tumors. However, variability in toxicity and response remains a major problem for patients receiving capecitabine. It is general that there are many factors for individual differences of drugs in clinical application, of which genetic factors accounted for more than 20%. Toxicities of capecitabine, such as diarrhea, hand-foot syndrome or anemia, were evaluated for possible relationship with pharmacogenetic polymorphisms in several pharmacogenomics studies. Due to the levels of evidence of those studies are low and lack of sufficient research data of Chinese, it has the important significance in studying individual differences of capecitabine in toxicities, through the pharmacogenomics research.

The aim of this study is to evaluating the association genetic polymorphisms with capecitabine-based chemotherapy toxicities in chinese solid tumor patients. By detecting the gene polymorphism, investigators intend to study the pharmacokinetic/pharmacogenomics (PK-PG) correlation of capecitabine and provide scientific basis for precise medication guide for people to use capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Any native Chinese men or women at least 18 years of age;
* Sign informed consent of the research;
* Have a histologic or cytologic diagnosis of solid tumor;
* Will receive capecitabine-based chemotherapy; Or patients who received capecitabine chemotherapy meet the inclusion and exclusion criteria of the research, and their clinical information is complete to obtain;
* Male and female patients with reproductive potential must use an approved contraceptive method during and for 3 months after discontinuation of study treatment.Women with childbearing potential must have a negative pregnancy test within 7 days prior to study enrollment;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Have discontinued all previous therapies for cancer for at least 28 days prior to study entry, and have recovered from the acute effects of therapy.
* Have adequate organ function, including:

  1. Bone marrow reserve:

     1. ANC≥1.5×109/L
     2. PLT≥100×109/L
     3. HGB≥10g/dL
  2. Hepatic:

     1. Bilirubin ≤ 1.5ULN
     2. ALT, AST ≤2.5 ULN, ≤5ULN when liver metastases are known.
  3. Renal: Src ≤1.5mg/dl
* Electrolytes: Patients may be entered into the study if, in the investigators' opinion, any electrolyte disorders, including K<3.4mEq/L, Ca<8.4mEq/L, or Mg<1.2mEq/l, may be appropriately managed and stabilized by the time of the laboratory evaluation prior to the chemotherapy. If electrolytes have not been stabilized during this time, the patient will be discontinued from the study.
* Have an estimated life expectancy, in the judgment of the investigator, which will permit the patient to complete the PK phase and at least 2 cycle of the evaluation of the toxicities.

Exclusion Criteria:

* Serious concomitant systemic disorder, including active infection, which is incompatible with the study (at the discretion of the investigator).
* History of human immunodeficiency virus, hepatitis B, or hepatitis C infections.
* Cardiac: Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV. It is recommended that patients with arrhythmias (persistent or paroxysmal ventricular or supraventricular arrhythmias, including atrial fibrillation or bradycardia (heart rate <50 beats per minute))be excluded at the investigator's discretion.
* Known family history of unexplained sudden death.
* Personal history of unexplained syncope within the last year.
* Patients with complete gastrectomy or other significant gastrointestinal diseases that, in the investigator's opinion, may significantly impact drug absorption.
* Inability to swallow tablets.
* Women who are breast feeding, lactating, or pregnant.
* Patients with known allergies to capecit and its supplementary materials.
* Drugs and herbal supplements that are known to be potent or moderate inhibitors or inducers of cytochrome P450 (CYP) are specifically excluded. Foods that are known to be potent or moderate inhibitors of CYP are also specifically excluded during the study.
* Patients receiving herbal regimens.
* Use of drugs with narrow therapeutic windows that are also known substrates of CYP2C9.
* Patients with DPYD deficiency.
* History of administration Usevir or its analogs within 28 days.
* Patients with severe renal impairment (CrCl <30ml/min)
* Failure for any reason to satisfy the investigator for adequate fitness to participated in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese solid tumor patients with the treatment of capecitabine-based chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe diarrhea toxicity | At 1 year
  The toxicity induced by capecitabine-based chemotherapy during observation time will be estimated on the basis of the National Cancer Institute Common Toxicity Criteria Version 4.03. Patients with grade 3-4 adverse events will be considered as having severe toxicity. At the end of each cycle (each cycle is 21 days) the grade will be scored. And the severest grade will be recorded and used for analysis.
Incidence of severe hand-foot syndrome toxicity | At 1 year
  The toxicity induced by capecitabine-based chemotherapy during observation time will be estimated on the basis of the National Cancer Institute Common Toxicity Criteria Version 4.03. Patients with grade 3-4 adverse events will be considered as having severe toxicity. At the end of each cycle (each cycle is 21 days) the grade will be scored. And the severest grade will be recorded and used for analysis.

SECONDARY OUTCOMES:
Incidence of other severe toxicities | At 1 year
  The other toxicities induced by capecitabine-based chemotherapy during observation time, including gastrointestinal toxicity, neurotoxicity, hematological toxicity etc., will be estimated on the basis of the National Cancer Institute Common Toxicity Criteria Version 4.03. Toxicities with grade 3-4 will be considered as severe toxicity, except for severe neurotoxicity (grade 2-3). At the end of each cycle (each cycle is 21 days) the grade will be scored. And the severest grade will be recorded and used for analysis.
Genotyping | Before chemotherapy
  Collect blood specimen, then detect genotype by next generation sequencing.
The kinds of the metabolites | Pre-dose and 3 hours after the last administration in the first cycle
  Determine the metabolic profiles of capecitabine. This outcome is not applicable to patients retrospectively collected.
Area under the curve [AUC] | Pre-dose and 3 hours after the last administration in the first cycle
  Determine the AUC of capecitabine and its metabolites. This outcome is not applicable to patients retrospectively collected.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality
  - Fuling Center Hospital of Chongqing City, Chongqing, Chongqing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Yunnan Cancer Hospital, Kunming, Yunnan